CLINICAL TRIAL: NCT04898621
Title: The Effect of Dietary Fructose on Gut Microbiota and Hepatosteatosis in Healthy Men
Brief Title: Dietary Fructose on Microbiota and Hepatosteatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Director, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZSE202105
Record Dates: First submitted 2021-05-14; First posted 2021-05-24 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hepatic Steatosis; Dietary Fructose Exposure
Keywords: Fructose; Microbiota; NAFLD
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: 60 healthy men will be recruited according to the inclusion criteria. All the participates are randomly allocated to Group A and Group B. Subjects in Group A will be instructed to drink fructose solution containing 75g fructose per day and those in Group B will be instructed to drink 150g fructose per day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subjects in Group A will drink 75g fructose solution daily for 4 weeks.
  Interventions: Dietary Supplement: 75g fructose solution
- Group B (Experimental): Subjects in Group B will drink 150g fructose solution daily for 4 weeks.
  Interventions: Dietary Supplement: 150g fructose solution

INTERVENTIONS:
Dietary Supplement: 75g fructose solution — Subjects will drink a bottle of 350 ml solution containing 75g fructose per day for 4 weeks.
  Arms: Group A
Dietary Supplement: 150g fructose solution — Subjects will drink a bottle of 700 ml solution containing 150g fructose per day for 4 weeks.
  Arms: Group B

SUMMARY:
The consumption of sugar-sweetened beverages (SSB) has increased steadily over the past decades, resulting in the dramatic increase of fructose intake as it is one of the main ingredients of artificial sweeteners. Recently, large epidemiological studies have documented the association between a high-fructose-diet and hepatic steatosis, and other metabolic disorders. So it is interesting for scientists to explore the underlying mechanism. This study aims to investigate the effect of dietary fructose and gut microbiota and the hepatosteatosis in healthy men. Serum and fecal metabolomics will be investigated.

DETAILED DESCRIPTION:
This is a single center, randomized, controlled study. 60 healthy men will be recruited according to the inclusion criteria. All subjects are randomly allocated to Group A and Group B, who orally takes 75g and 150g fructose daily respectively. Subjects in Group A will be instructed to drink fructose solution containing 75g fructose per day, and those in Group B will be instructed to drink fructose solution containing 150g fructose per day. The intervention will last four weeks. The anthropomentric data will be collect with questionnaire and serum and fecal samples collected at baseline and the end of the intervention. The effect and mutual interaction of dietary fructose and microbiota will be explored. The effect of dietary fructose on hepatosteatosis will be investigated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged from 18 to 40 (including both ends);
2. Body mass index (BMI) ranges from 18.5 to 23.9 kg/m2 (including both ends);
3. The body weight has not changed dramatically in the past 3 months (±3kg);

Exclusion Criteria:

1. Subjects who have received antibiotic-related treatment, proton pump inhibitor treatment, or glucocorticoid hormone treatment within 1 month before enrollment;
2. Subjects with diabetes or cardiovascular disease or other chronic diseases who require long-term medication;
3. Subjects who suffered from an acute gastrointestinal diseases within the past month, or who have an history of chronic gastrointestinal disease or hepatitis;
4. Subjects with a history of gastrointestinal surgery;
5. Subjects with abnormal liver or kidney function, or severe cardiovascular diseases;
6. Subjects with mental disorders or impaired cognitive function;
7. Poor compliance;
8. Participates enrolled in other clinical research at the same time;
9. Other unsuitable occasions judged by clinicians..

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of microbiota | 4 weeks
  The change of microbiota in fecal samples from baseline to the end of the study
Change of intra-hepatic triglyceride content(IHTG) | 4 weeks
  The IHTG will be measured using MRI-PDFF

SECONDARY OUTCOMES:
Change of serum metabolomics | 4 weeks
  Serum metabolomics will be determined using MS.
The change of serum proinflammatory factors | 4 weeks
  Serum proinflammatory factors, including TNFa, IL-6 will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Endocrinology, Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Li Y, Teng D, Shi X, Qin G, Qin Y, Quan H, Shi B, Sun H, Ba J, Chen B, Du J, He L, Lai X, Li Y, Chi H, Liao E, Liu C, Liu L, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Teng W, Shan Z. Prevalence of diabetes recorded in mainland China using 2018 diagnostic criteria from the American Diabetes Association: national cross sectional study. BMJ. 2020 Apr 28;369:m997. doi: 10.1136/bmj.m997. PMID 32345662
- [Background] Samuel VT, Shulman GI. Nonalcoholic Fatty Liver Disease as a Nexus of Metabolic and Hepatic Diseases. Cell Metab. 2018 Jan 9;27(1):22-41. doi: 10.1016/j.cmet.2017.08.002. Epub 2017 Aug 31. PMID 28867301
- [Background] Bray GA, Nielsen SJ, Popkin BM. Consumption of high-fructose corn syrup in beverages may play a role in the epidemic of obesity. Am J Clin Nutr. 2004 Apr;79(4):537-43. doi: 10.1093/ajcn/79.4.537. PMID 15051594
- [Background] Zhao S, Jang C, Liu J, Uehara K, Gilbert M, Izzo L, Zeng X, Trefely S, Fernandez S, Carrer A, Miller KD, Schug ZT, Snyder NW, Gade TP, Titchenell PM, Rabinowitz JD, Wellen KE. Dietary fructose feeds hepatic lipogenesis via microbiota-derived acetate. Nature. 2020 Mar;579(7800):586-591. doi: 10.1038/s41586-020-2101-7. Epub 2020 Mar 18. PMID 32214246
- [Background] Hugenholtz F, de Vos WM. Mouse models for human intestinal microbiota research: a critical evaluation. Cell Mol Life Sci. 2018 Jan;75(1):149-160. doi: 10.1007/s00018-017-2693-8. Epub 2017 Nov 9. PMID 29124307
- [Background] Jensen T, Abdelmalek MF, Sullivan S, Nadeau KJ, Green M, Roncal C, Nakagawa T, Kuwabara M, Sato Y, Kang DH, Tolan DR, Sanchez-Lozada LG, Rosen HR, Lanaspa MA, Diehl AM, Johnson RJ. Fructose and sugar: A major mediator of non-alcoholic fatty liver disease. J Hepatol. 2018 May;68(5):1063-1075. doi: 10.1016/j.jhep.2018.01.019. Epub 2018 Feb 2. PMID 29408694
- [Background] Taskinen MR, Soderlund S, Bogl LH, Hakkarainen A, Matikainen N, Pietilainen KH, Rasanen S, Lundbom N, Bjornson E, Eliasson B, Mancina RM, Romeo S, Almeras N, Pepa GD, Vetrani C, Prinster A, Annuzzi G, Rivellese A, Despres JP, Boren J. Adverse effects of fructose on cardiometabolic risk factors and hepatic lipid metabolism in subjects with abdominal obesity. J Intern Med. 2017 Aug;282(2):187-201. doi: 10.1111/joim.12632. Epub 2017 Jun 27. PMID 28548281
- [Background] Silbernagel G, Machann J, Unmuth S, Schick F, Stefan N, Haring HU, Fritsche A. Effects of 4-week very-high-fructose/glucose diets on insulin sensitivity, visceral fat and intrahepatic lipids: an exploratory trial. Br J Nutr. 2011 Jul;106(1):79-86. doi: 10.1017/S000711451000574X. Epub 2011 Mar 14. PMID 21396140
- [Background] Smajis S, Gajdosik M, Pfleger L, Traussnigg S, Kienbacher C, Halilbasic E, Ranzenberger-Haider T, Stangl A, Beiglbock H, Wolf P, Lamp T, Hofer A, Gastaldelli A, Barbieri C, Luger A, Trattnig S, Kautzky-Willer A, Krssak M, Trauner M, Krebs M. Metabolic effects of a prolonged, very-high-dose dietary fructose challenge in healthy subjects. Am J Clin Nutr. 2020 Feb 1;111(2):369-377. doi: 10.1093/ajcn/nqz271. PMID 31796953
- [Background] Teff KL, Grudziak J, Townsend RR, Dunn TN, Grant RW, Adams SH, Keim NL, Cummings BP, Stanhope KL, Havel PJ. Endocrine and metabolic effects of consuming fructose- and glucose-sweetened beverages with meals in obese men and women: influence of insulin resistance on plasma triglyceride responses. J Clin Endocrinol Metab. 2009 May;94(5):1562-9. doi: 10.1210/jc.2008-2192. Epub 2009 Feb 10. PMID 19208729
- [Background] Blaak E. Gender differences in fat metabolism. Curr Opin Clin Nutr Metab Care. 2001 Nov;4(6):499-502. doi: 10.1097/00075197-200111000-00006. PMID 11706283
- [Background] Mosca L, Barrett-Connor E, Wenger NK. Sex/gender differences in cardiovascular disease prevention: what a difference a decade makes. Circulation. 2011 Nov 8;124(19):2145-54. doi: 10.1161/CIRCULATIONAHA.110.968792. PMID 22064958
- [Background] Karlsson FH, Nookaew I, Nielsen J. Metagenomic data utilization and analysis (MEDUSA) and construction of a global gut microbial gene catalogue. PLoS Comput Biol. 2014 Jul 10;10(7):e1003706. doi: 10.1371/journal.pcbi.1003706. eCollection 2014 Jul. PMID 25010449
- [Background] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281